CLINICAL TRIAL: NCT04687007
Title: SMART-ALD - A New Lifestyle Intervention to Improve Physical and Mental Well-being and Quality of Life in Women With X-linked Adrenoleukodystrophy (X-ALD)
Brief Title: SMART-ALD - A New Lifestyle Intervention to Improve Quality of Life in Women With X-linked Adrenoleukodystrophy (X-ALD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leipzig University Medical Center (Other)
Collaborators: European Leukodystrophy Association (Other)
Responsible Party: Principal Investigator, Lisa Schäfer, Dr., Leipzig University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ELA FOA2020-002
Record Dates: First submitted 2020-12-11; First posted 2020-12-29 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: Adrenoleukodystrophy; Adrenomyeloneuropathy; Genetic Diseases, X-Linked; Rare White Matter Disorders; Female Carriers; Women with X-ALD; Peroxisomal Disorders; eHealth Intervention; Central Nervous System Diseases; Heterozygous Carriers; Quality of Life; Lifestyle Intervention
MeSH Terms: conditions — Adrenoleukodystrophy; Genetic Diseases, X-Linked; Peroxisomal Disorders; Central Nervous System Diseases | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 12 months of SMART-ALD intervention (experimental group; EG) or a waiting list control group (CG), in which patients receive 6 months of SMART-ALD after a 6-months waiting period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART-ALD - Experimental group (EG) (Experimental): Participants will receive 12 months of SMART-ALD intervention
  Interventions: Behavioral: SMART-ALD
- Waiting List - Control group (CG) (Other): Participants will receive 6 months of SMART-ALD after a 6-months waiting period
  Interventions: Behavioral: Waiting list

INTERVENTIONS:
Behavioral: SMART-ALD — At the beginning of SMART-ALD, a multi-professional team evaluates participant's current health status and develops an individual treatment plan together with the participant. The SMART-ALD intervention offers medical, psychological, and social counseling, as well as a physical fitness and disease-specific nutritional program carried out via video consultation. Thus, scope and intensity of SMART-ALD intervention is initially tailored to individual needs and continuously adapted to changes during intervention.
  Arms: SMART-ALD - Experimental group (EG)
Behavioral: Waiting list — At the beginning of the study, patients of the waiting list (WL) control condition receive one medical consultation via video consultation, including recommendations to contact their local treating physician if necessary. Individuals are instructed not to seek any other medical or psychological treatment for X-ALD symptoms without informing the study staff. All WL patients are guaranteed 6 months of SMART-ALD intervention after a waiting period of 6 months.
  Arms: Waiting List - Control group (CG)

SUMMARY:
X-linked Adrenoleukodystrophy (X-ALD) is one of the most frequent inborn error of metabolism caused by mutations in the ABCD1 gene, which codes for the transporter of saturated very long-chain fatty acids (VLCFA) for peroxisomal degradation, thus causing their toxic accumulation in body fluids and tissues. The clinical spectrum ranges from adrenal insufficiency without neurological symptoms to a rapidly progressive, fatal cerebral demyelinating disease that may occur in childhood as well as later in life. The most frequent phenotype in adulthood is adrenomyeloneuropathy (AMN), a slowly progressive myelopathy and peripheral neuropathy, which may also be prevalent in up to 80% of females carrying the X-ALD gene defect. Since signs and symptoms in females are usually milder and with a later onset, they are frequently underestimated, overlooked or misinterpreted, e.g. as Multiple Sclerosis. Consequently, many women with X-ALD do not receive adequate treatment.

Against this background, the development of new therapeutic interventions with the help of eHealth technology (e.g., counselling and treatment via digital communication tools) is of particular relevance, as it provides cost-effective, regular care even for patients who live remote from Leukodystrophy clinics.

The aims of this study is to evaluate the effectiveness of a multi-approach intervention ("SMART-ALD") on physical and mental well-being and quality of life in n=30 X-ALD symptomatic heterozygous females compared to a waiting list control group (n=30) using electronic health (ehealth) technology.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the patient or a competent guardian with legal capacity to execute a local Institutional Review Board/Independent Ethics Committee approved consent.
* Females ≥18 years at the time of consent, with proven X-ALD as defined by

  1. Elevated VLCFA values, or
  2. Mutation in ABCD1 gene
* Neurological symptoms as defined by Adult ALD Clinical Score (AACS) ≥ 2

Exclusion Criteria:

* No informed consent and assent
* Any medical condition that may interfere with the study, e.g. severe liver, kidney, active infections or major heart diseases (>New York Heart Association class II)
* Any clinically significant condition with an estimated life-expectancy of <6 months
* Current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported quality of life (assessed via Short Form Health Survey, SF-36; range: 0-100, with higher scores indicating better quality of life) 6 months after randomization (=after 6 months SMART-ALD) in the EG compared to waiting list CG | 6 months

SECONDARY OUTCOMES:
Changes in objectively measured neurological symptoms (Adult Adrenoleukodystrophy Clinical Score, AACS; range: 0-24, with higher scores indicating greater impairment) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in motor functions (objectively measured via timed 25-foot walk test, T25FW) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in objectively measured activity index (pedometer - fitness tracker wrist band) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in self-reported functional status (assessed via Activity of Daily Living Score, ADLs, range: 0-6, with higher scores indicating better functioning) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in self-reported mental health (Beck Depression Inventory, BDI-II, range: 0-63, with higher scores indicating greater depression) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in self-reported chronic pain (Brief Pain Inventory, BPI, range: 0-10, with higher scores indicating greater pain) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in self-reported sleep quality (Pittsburgh Sleep Quality Index, PSQI, range: 0-21, with higher scores indicating worse sleep quality) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in self-reported fatigue symptoms (Modified Fatigue Impact Scale, MFIS, range: 0-84, with higher scores indicating greater fatigue) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months
Changes in self-reported sexual functionality (Female Sexual Function Index, FSFI, range: 2-36, with higher scores indicating better sexual function) 6 and 12 months after randomization in the EG compared to waiting list CG | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Köhler, MD, Principal Investigator — Leipzig University Medical Center, Leukodystrophy Outpatient Clinic, Department of Neurology, Leipzig, Germany
Locations (2):
- Germany (2):
  - Leipzig University Medical Center, Leukodystrophy Outpatient Clinic, Department of Neurology, Leipzig, Germany, Leipzig, Saxony
  - Leukodystrophy Outpatient Clinic, Leipzig

REFERENCES:
- [Derived] Schafer L, Unterlauft A, Froebrich-Andress B, Wollny C, Rossler M, Fischer R, Bahr C, Lier J, Wasmus DT, Bergner CC, Kohler W. Improving quality of life in rare diseases using disease-specific, multidisciplinary online interventions on the example of rare X-linked adrenoleukodystrophy: a randomized-controlled trial. Ther Adv Neurol Disord. 2025 Sep 28;18:17562864251376109. doi: 10.1177/17562864251376109. eCollection 2025. PMID 41030609